CLINICAL TRIAL: NCT01472458
Title: Premature Termination of Resuscitation in Survivors of Cardiac Arrest
Acronym: PremaTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Damon Scales, Scientist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: SPARC - PremaTOR
Record Dates: First submitted 2011-08-02; First posted 2011-11-16 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Hypothermia; Post Cardiac Arrest Care; Survivors of cardiac arrest
MeSH Terms: conditions — Heart Arrest; Hypothermia | interventions — Quality Improvement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Intervention (Active Comparator): This stepped-wedge cluster randomized evaluation will randomly allocate 18 hospitals into 4 groups to receive our active intervention at different sequential time points according to the randomly assigned stepped-wedge schedule. Hospitals will function as control hospitals until it is their turn to receive the active intervention, according to the stepped wedge schedule. Each wedge consists of 4-5 hospitals and will last 5 months.
  Interventions: Behavioral: Quality improvement
- Control Hospitals (No Intervention): This stepped-wedge cluster randomized evaluation will randomly allocate 18 hospitals into 4 groups to receive our active intervention at different sequential time points according to the randomly assigned stepped-wedge schedule. Hospitals will function as control hospitals until it is their turn to receive the active intervention, according to the stepped wedge schedule. Each wedge consists of 4-5 hospitals and will last 5 months.

INTERVENTIONS:
Behavioral: Quality improvement — The primary intervention in this project will be a multi-faceted quality improvement plan targeting improved predictions of neurological outcome and survival after cardiac arrest.
  Arms: Active Intervention

SUMMARY:
The study Premature Termination of Resuscitation in Survivors of Cardiac Arrest focuses on using innovative knowledge translation strategies to improve appropriate neuroprognostication for survivors of cardiac arrest and prevent premature termination of life sustaining therapies. This is important because any early gains achieved during resuscitation will be nullified if clinicians terminate life-sustaining therapies prematurely based on inadequate prognostic information. An effective translation strategy for neuroprognostication will result in improved physician adherence to evidence-based medicine and an increase in the proportion of patients surviving to achieve a good neurological outcome following cardiac arrest.

DETAILED DESCRIPTION:
A stepped wedge cluster randomized trial design will be employed in order to properly evaluate the impact of this intervention. Each of the 18 participating hospitals will be randomized one of the four wedges according to a random schedule; each wedge will consist of 4 to 5 hospitals. With this design, the implementation of the intervention will be rolled out sequentially to the participating hospitals over a 5 month period for each wedge. All hospitals will have received the intervention by the end of the study.

Note that the study design fields provided by ClinicalTrials.gov do not allow for describing this type of study design; therefore, the investigators have listed the study as a single arm. In reality, this study will have 4 wedges, each containing randomized clusters of 4-5 hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients =/> 18 years of age
* Non-traumatic out of hospital cardiac arrest
* Sustained return of spontaneous circulation (palpable pulse for > 20 minutes)
* Comatose (i.e. without full neurological recovery; non-responsive to verbal commands)
* Surviving to at least 6 hours after emergency department arrival

Exclusion Criteria:

* Patients who die within 6 hours of emergency department arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2011-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Effective knowledge strategy | Two years
  Our primary endpoint measures the uptake of appropriate neurological prognostication in survivors of cardiac arrest. We define appropriate neurological prognostication as the number of patients that have appropriate prognostic testing (as recommended by Advanced Life Support/ILCOR guidelines) performed before death but occurring at least 72 hours after the cardiac arrest; the denominator for this endpoint is the total number of patients admitted to hospital following cardiac arrest excluding deaths unrelated to predictions of poor neurological prognosis.

SECONDARY OUTCOMES:
Qualitative Aim | Two years
  To understand reasons for premature termination of life sustaining therapy and barriers to evidence based neurological prognostication in survivors of cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Damon C Scales, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre

REFERENCES:
- [Derived] Scales DC, Golan E, Pinto R, Brooks SC, Chapman M, Dale CM, Jichici D, Rubenfeld GD, Morrison LJ; Strategies for Post-Arrest Resuscitation Care Network. Improving Appropriate Neurologic Prognostication after Cardiac Arrest. A Stepped Wedge Cluster Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Nov 1;194(9):1083-1091. doi: 10.1164/rccm.201602-0397OC. PMID 27115286